CLINICAL TRIAL: NCT02078115
Title: Observational Study of Blood Pressure Control Pattern and the Impact on the Target Organ Damages
Brief Title: Assessment of Blood Pressure Control and Target Organ Damage in Patients With Chronic Kidney Disease and Hypertension -II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yon Su Kim, Professor, Seoul National University Hospital
Other Study IDs: APRODITE-2; Boryung (Other Grant/Funding Number: Boryung)
Record Dates: First submitted 2014-02-05; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Disease; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic kidney disease, hypertension: 20 <= age < 75 years 15 <= estimated glomerular filtration rate (GFR) < 90

SUMMARY:
The purpose of this study is to find the change of blood pressure (BP) control pattern (true controlled, white-coat, masked, and sustained uncontrolled/ dipper, non-dipper, reverse-dipper, and extreme-dipper) in patients with chronic kidney disease (CKD) over 3 years. And Other objective is the relationship between the BP control pattern and the target organ damages such as renal function, proteinuria, left ventricular hypertrophy (LVH), and so on. In addition, we will find clinical factors related to the BP control pattern.

ELIGIBILITY:
Inclusion Criteria:

1. with informed consent
2. 20 <= age < 75 years
3. diagnosed as hypertension 6 months (or 3 visits) prior to enrollment, taking anti-hypertensive drugs over 3 months
4. all-cause chronic kidney disease patients with 15 <= estimated GFR < 90
5. no change of anti-hypertensive drugs within 2 weeks and good compliance

Exclusion Criteria:

1. changed prescription according to ambulatory blood pressure monitoring (ABPM) regularly
2. had acute kidney injury/hospitalization
3. had a proteinuria of > 6 g/day (spot urine protein to creatinine ratio > 6.0 g/g Cr)
4. had end stage renal disease (ESRD) with dialysis and/or were a kidney recipient
5. had diseases, such as uncontrolled arrhythmia, uncontrolled bronchial asthma/chronic obstructive pulmonary disease, or primary endocrinologic diseases except diabetes mellitus
6. were pregnant/lactating women
7. were night shift workers.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic kidney disease patients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The change of blood pressure control pattern in patients with CKD | 1 year after enrolling the last participant

SECONDARY OUTCOMES:
1) target organ damages in kidney and heart | 1 year after enrolling the last participant
2) the relationship between the change of BP control pattern and the target organ damages | 1 year after enrolling the last participant
3) assessment of related clinical factors with BP control pattern | 1 year after enrolling the last participant

CONTACTS AND LOCATIONS:
Overall Officials: Sung Kyun Kim, MD, Study Director — Hallym University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea